CLINICAL TRIAL: NCT01116258
Title: A Phase I, Single-center, Double-blind, Randomized, Placebo-controlled, Parallel-group, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD5847 Following Oral Administration to Healthy Male Subjects and Female Subjects of Non-childbearing Potential
Brief Title: A Study in Healthy Volunteers to Assess Safety and Blood Levels of AZD5847 After Multiple Doses Over 14 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3430C00002
Record Dates: First submitted 2010-04-29; First posted 2010-05-04 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Safety
MeSH Terms: interventions — posizolid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD5847
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5847 — oral suspension, 15 days
  Arms: 1
Drug: Placebo — oral suspension, 15 days
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety, tolerability and blood levels of AZD5847 after daily oral dosing for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18-30

Exclusion Criteria:

* Use of drugs that inhibit or induce cytochrome P450 3A4 enzymes
* History of presence of gastrointestinal, hepatic or renal disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, vital signs, physical examinations, clinical laboratory assessments, 12-lead ECG, digital ECG, telemetry) | collected prior to treatment, during treatment, and follow-up for a total of 25 to 52 days(includes upto 28 days for screening)

SECONDARY OUTCOMES:
characterize the Pharmacokinetics of AZD9742 in blood and urine | PK-sampling during 14 pre-defined study days for PK profiling

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shaw, Study Director — AstraZeneca; Brendan Smyth, Study Chair — AstraZeneca; David Melnick, Study Director — AstraZeneca; Eleanor Lisbon, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Overland Park, Kansas, United States